CLINICAL TRIAL: NCT06934746
Title: Evaluation of Screen Time and Digital Media on ADHD
Acronym: ADHD
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Janice Gamil Sadek Zakka, Resident of pediatric, Assiut University
Other Study IDs: role of digital media in ADHD
Record Dates: First submitted 2025-04-06; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Monitor Adverse Events

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 130 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: DSM-5 criteria. — The DSM-5 defines three levels of ADHD severity based on symptom count and frequency: 1. Mild ADHD • Symptom Count: Just meets the diagnostic criteria (6 symptoms in children for either inattention or hyperactivity/impulsivity). • Frequency: Symptoms occur but are not excessively frequent. 2. Moderate ADHD • Symptom Count: More than the minimum required for diagnosis. • Frequency: Symptoms occur frequently (e.g., several times a week). 3. Severe ADHD • Symptom Count: Many symptoms well beyond the diagnostic threshold. • Frequency: Symptoms occur daily or multiple times per day.(National Center for Biotechnology Information, n.d.)

SUMMARY:
1. Assess how different types of digital media influence inattention, impulsivity, and hyperactivity in children with ADHD.
2. Analyze the role of screen time duration, content type, parental supervision, and socioeconomic status in ADHD symptom severity.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is one of the most prevalent neurodevelopmental disorders in children, characterized by persistent patterns of inattention, hyperactivity, and impulsivity. Studies suggest that its prevalence has risen due to improved recognition and changing diagnostic criteria. Children with ADHD experience significant challenges in school performance, including difficulty sustaining attention, frequent careless mistakes, and trouble following instructions, all of which contribute to lower academic achievement and increased need for special education support. ADHD is linked to problematic eating behaviors, as irregular meal patterns, increased consumption of unhealthy foods, and a higher risk of obesity due to impulsivity and poor self-regulation. Beyond academics and nutrition, ADHD also affects sleep quality, emotional regulation, and social interactions, leading to increased behavioral issues and conflicts with peers and family members. The widespread use of digital media further complicates these challenges, as excessive screen time has been associated with exacerbating ADHD symptoms and negatively impacting cognitive and emotional development. These findings highlight the urgent need for targeted interventions to support children with ADHD across multiple aspects of their daily lives

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed children with ADHD, confirmed by DSM-5 and Gilliam ADHD rating scale. • Parental consent for participation.

Exclusion Criteria:

* Comorbid neurodevelopmental disorders (e.g., autism, intellectual disability). • Chronic medical conditions affecting cognitive or behavioral function.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neuro-psychiatric Outpatient clinic in Assiut University Children Hospita
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Inattention Symptoms Measured by the ADHD Rating Scale-IV | Baseline (Day 1) and after 6 months of follow-up
  Evaluate the change in inattention symptoms before and after exposure to different types of digital media (e.g., videos, games, educational apps) using the ADHD Rating Scale-IV completed by parents or caregivers.
Change in Hyperactivity/Impulsivity Symptoms Measured by the ADHD Rating Scale-IV | Baseline (Day 1) and after 6 months of follow-up
  Assess the change in hyperactivity and impulsivity symptoms in children with ADHD in relation to total daily screen time, content type, and level of parental supervision, using the ADHD Rating Scale-IV.

SECONDARY OUTCOMES:
Correlation between Socioeconomic Status and ADHD Symptom Severity | After 6 months of follow-up
  Analyze the association between family socioeconomic status (SES) and the severity of ADHD symptoms after 6 months of exposure to digital media, using standardized SES assessment tools and ADHD Rating Scale-IV scores.